CLINICAL TRIAL: NCT01376193
Title: Drug Use Investigation for AMERGE (Naratriptan Hydrochloride) Tablet
Status: Completed | Type: Observational
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Other Study IDs: 112924
Record Dates: First submitted 2011-06-09; First posted 2011-06-20 (Estimated); Last update posted 2013-05-20 (Estimated); Status verified 2013-05

CONDITIONS: Migraine Disorders
MeSH Terms: conditions — Migraine Disorders | interventions — naratriptan

STUDY DESIGN:
Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Subjects prescribed naratriptan tablets: Subjects with migraine headache prescribed naratriptan tablets during study period
  Interventions: Drug: Naratriptan

INTERVENTIONS:
Drug: Naratriptan — Collection of safety data

SUMMARY:
The study is designed to investigate the information on safety and efficacy of naratriptan tablets on Japanese subjects with migraine headache during Japanese post-marketing surveillance period.

ELIGIBILITY:
Inclusion Criteria:

* Subjects with migraine headache
* Must use naratriptan tablets for the first time

Exclusion Criteria:

* Subjects with hypersensitivity to naratriptan
* Subjects with history, symptoms, or signs of myocardial infarction, ischemic cardiac disease, or variant angina
* Subjects with history of peripheral vascular disorder
* Subjects with history of cerebrovascular disorder or transient ischemic attacks
* Subjects with uncontrolled high-blood pressure
* Subjects with severe hepatic function disorder or renal function disorder
* Subjects taking ergotamine, ergotamine derivative containing product, or 5-HT1B/1D agonist

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Japanese subjects with migraine headache
Sampling Method: Probability Sample
Enrollment: 500 (Actual)
Dates: Start 2009-04; Primary Completion 2011-10 (Actual); Study Completion 2011-10 (Actual)

PRIMARY OUTCOMES:
The number of incidence of adverse events in subjects with migraine headache | 2 months

SECONDARY OUTCOMES:
Occurrence of cardiovascular-related adverse events | 2 months
  Occurrence of cardiovascular-related adverse events is investigated throughout study period
Occurrence of cerebrovascular disorder | 2 months
  Occurrence of cerebrovascular disorder is investigated throughout study period
Occurrence of serotonin syndrome | 2 months
  Occurrence of serotonin syndrome is investigated throughout study period

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline

REFERENCES:
- [Background] Takao Takeshima, Atsuko Ishida, Terufumi Hara. Drug Use Investigation on Naratriptan Tablets (Amerge®) in Patients with Migraine. [Prog Med]. 2012;32(8):95-105.